CLINICAL TRIAL: NCT01237834
Title: Physiological Responses in Tobacco Chippers (Non Nicotine-dependent Light Smokers)
Brief Title: Physiological Responses in Tobacco Chippers
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Barry S. Oken, MD, Oregon Health and Science University
Other Study IDs: IRB6698
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Smoking; Stress
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Heavy smokers, 15 or more cigarettes/day: Nicotine dependent.
- Light smokers (chippers): Less than 2 cigarettes/day, at least 2 days/week. Non nicotine-dependent.
- Non smokers

SUMMARY:
This study will analyze a series of biological and behavioral markers in different populations of smokers. The study groups will differ in their cigarette consumption and level of nicotine dependence. This analysis will help to identify factors that might be important for smoking behavior and nicotine addiction. The results from this study will contribute to improve campaigns for smoking prevention and treatments for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* age 25-55

Exclusion Criteria:

* alcohol or drug addiction
* unstable significant medical problems
* neurologic disease
* medications known to affect CNS function or impact physiologic parameters measured in the study
* significant visual impairment
* breath carbon monoxide (BCO) level of less than 10 ppm for smokers
* breath carbon monoxide (BCO) level of more than 5 ppm for non-smokers
* for heavy regular smokers: erratic smoking history (i.e. they must have smoked an average of 15 cigarettes daily for at least one year)

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Electroencephalography | Changes from baseline during a hard cognitive task
  Electroencephalography will be measured during performance on a hard cognitive task.

SECONDARY OUTCOMES:
Salivary cortisol | Changes from baseline during performance on a hard cognitive task
  Salivary cortisol will be measured at baseline, during a hard cognitive task and 30 minutes after the cognitive task.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Oken, Principal Investigator — Oregon Health and Science University; Laura Carim Todd, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States